CLINICAL TRIAL: NCT04054622
Title: Patient-ventilator Asychrony During Non-invasive Ventilation When COPD Patients Doing Exercise
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenfeng He, Principle investigator, Guangzhou Medical University
Other Study IDs: GIRH-201922
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: COP; Non-invasive Ventilation; Pulmonary Rehabilitation
Keywords: patient-ventilator asynchrony
MeSH Terms: conditions — Patient-Ventilator Asynchrony

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary rehabilitation programmes including aerobic exercise training have strong evidence of effectiveness in improving exercise capacity, dyspnoea and HRQL in patients with COPD. Therefore, current guidelines recommend pulmonary rehabilitation, including exercise training, in these patients. Non-invasive ventilation(NIV) is increasingly used during exercise training programmes in order to train patients at intensity levels higher than allowed by their clinical and pathophysiological conditions. Patient-ventilator asynchrony (PVA) describes the poor interaction between the patient and the ventilator and is the consequence of the respiratory muscle activity of the patient being opposed to the action of the ventilator.PVA have unfavourable clinical impace on gas exchange, dyspnoea perception, patient comfort and tolerance and reduced adherence to NIV. This study is going to detect whether the PVA will increase when COPD patients exercise with NIV supporingt

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80, males and females;
2. Stage III and IV COPD;
3. Similar with non-invasive ventilation;
4. Willing to participate in the study;
5. Able to provide informed consent.

Exclusion Criteria:

1. Presented with an acute exacerbation during previous 3 months;
2. Bronchiectasis; post-tuberculosis sequelae; rib cage deformities; neuromuscular disorders; and bronchial carcinoma.
3. Intolerant with NIV

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD, according to the criteria set by the Global Initiative for Obstructive Lung Disease scientific committee, were asked to participate in the present study. Patients had to meet the following inclusion criteria: 1) Age 40-80, males and females; 2) Stage III and IV COPD; 3) Similar with non-invasive ventilation; 4) Willing to participate in the study; 5) Able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Asynchrony index | 5 hours
  Asynchrony index is defined as the number of asynchrony events divided by the total respiratory rate computed as the sum of the number of ventilator cycles (triggered or not) and of wasted efforts: asynchrony Index (expressed in percentage) = number of asynchrony events/total respiratory rate (ventilator cycles +wasted efforts) × 100

SECONDARY OUTCOMES:
Severe Respiratory Insufficiency (SRI) Questionnaire | 5 hours
  The SRI Questionnaire has good psychometric properties shown to be valid for chronic hypercapnic COPD patients receiving NIV. It includes 49 items on seven subscales.
COPD assessment test | 5 hours
  The COPD Assessment Test is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time.
Partial pressure of arterial blood carbon dioxide (PaCO2) | 5 hours
  Daytime arterial blood gas samples were taken with patients resting in a sitting position and breathing room air without having used NIV for at least 1 hour.
6-minute walk test | 5 hours
  The 6-minute walk test plays a key role in evaluating functional exercise capacity, assessing prognosis and evaluating response to treatment across a wide range of respiratory diseases

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD, Study Director — Guangzhou Institute of Respiratory Health
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University., Guangzhou, Guangdong, China